CLINICAL TRIAL: NCT04322305
Title: A Double-blind, Placebo-Controlled Trial of Pregabalin for the Treatment of Alcohol Use Disorder
Brief Title: Pregabalin Trial for the Treatment of Alcohol Use Disorder
Acronym: GABI2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, John Mariani MD, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7977; R21AA028371 (NIH)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; treatment; pregabalin
MeSH Terms: conditions — Alcoholism | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Randomized Double blind, placebo controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Pregabalin will be administered in 75 mg and 100 capsules; placebo capsules will appear identical to the pregabalin capsules. Participants in both study arms will receive the same number of capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pregabalin (Experimental): Treatment with pregabalin administered in 75 mg and 100 capsules in dosages up to 600 mg per day for up to 8 weeks (including a 3 week titration run up) followed by a one week taper.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Individuals will receive the placebo capsules that appear identical to the pregabalin capsules and will receive the same number of capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin will be provided in 75 and 100 mg capsules twice daily for a maximum dose of 600 mg/day or the maximum tolerated dose over the 8 week medication phase and followed by a one week taper.
  Other Names: Lyrica
  Arms: Pregabalin
Other: Placebo — Placebo capsules will be provided twice daily over 8 weeks and one week taper..
  Arms: Placebo

SUMMARY:
In a 10-week randomized double-blind placebo-controlled outpatient pilot trial the efficacy of pregabalin in the treatment of alcohol dependence will be studied in 50 treatment-seeking outpatients. Participants will report drinking a minimum of 5 standard drinks for men or 4 standard drinks for women at least 4 days per week over the past 28 days.

DETAILED DESCRIPTION:
In a 10-week double-blind placebo controlled outpatient clinical trial, the safety and efficacy ofpregabalin will be tested in 50 outpatients with Alcohol Use Disorder.Participants will be randomly allocated (1:1) to receive pregabalin or an identical-appearing, inert placebo. All study medication (placebo and pregabalin) will be over-capsulated with riboflavin to assess compliance. Pregabalin will be administered in 75 mg and 100 capsules; placebo capsules will appear identical to the pregabalin capsules. Participants in both study arms will receive the same number of capsules. Pregabalin will be titrated over a 3-week period to the FDA maximum (600 mg per day) or the maximum tolerated dose.

Study visits will occur daily for the first 4 days of the study period, then approximately every other day for the remainder of week 1, for a total of 5 study visits (study days 1,2,3,4, and 5 or 7). During the second week, study visits will continue every other day for a total of 3 study visits (study days 8,10, and 12). During the remainder of the 8-week medication study period, study visits will occur twice weekly. There will be two visits during a post-study taper week (week 9) and a follow-up visit during week 10. One visit per week will be with the research psychiatrist. All participants will have a weekly supportive behavioral treatment session with the research psychiatrist using a manual designed for pharmacotherapy trials in subjects with alcohol use disorders

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 criteria for current alcohol use disorder
* Reports drinking a minimum of 5 standard drinks for men or 4 standard drinks for women at least 4 days per week over the past 28 days
* Between the ages of 18 and 65
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Subjects with any current psychiatric disorder as defined by DSM-5, other than Alcohol use disorder, that in the investigator's judgment likely requiring ongoing dosage adjustments of their current medications or requiring changes in their medication and/or might require intervention over the course of the study, including schizophrenia, schizoaffective disorder, psychotic disorders other than transient psychosis due to drug abuse, bipolar disorder, and current suicidality with plan and intent. Individuals who are currently stable on a psychotropic medication for at least 3 months may be included if in the investigator's opinion the psychotropic medication is compatible with the study medication (pregabalin). The medications being allowed are commonly used antidepressants, including the SSRIs (e.g., fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, escitalopram), SNRI's (e.g., venlafaxine, desvenlafaxine, duloxetine), and bupropion.
* Evidence of moderate-to-severe alcohol withdrawal Clinical Institute Withdrawal Assessment (revised version) (CIWA-Ar score ≥10)
* History of alcohol withdrawal seizures or alcohol withdrawal delirium
* History of allergic reaction to candidate medication (pregabalin)
* Pregnancy, lactation, or failure in female patients to use adequate contraceptive methods
* Unstable physical disorders which might make participation hazardous
* Subjects who have a current DSM-5 diagnosis of moderate or severe substance use disorder, with the exception of alcohol, nicotine and caffeine dependence. A diagnosis of a mild substance use disorder will not be exclusionary, as long as the current primary substance use disorder is alcohol dependence.
* Are legally mandated to participate in alcohol use disorder treatment program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of heavy drinking days | measured weekly over the 8 weeks of the medication phase of the trial or length of each individual's participation
  Change in heavy drinking days as quantified by the proportion of heavy drinking days (defined as any day where the number of standard drinks was at least 5 for men and at least 4 for women) per week as measured by the timeline follow-back (TLFB) method.

CONTACTS AND LOCATIONS:
Overall Officials: john mariani, MD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- Nyspi-Stars, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 12 months and ending 5 years after article publication
Access Criteria: to researcher who provides a methodologically sound proposal to achieve aims in the approved proposal